CLINICAL TRIAL: NCT03191292
Title: Bacterial Epidemiology and Empirical Antibiotherapy in Patients With Prosthetic Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0306
Record Dates: First submitted 2017-04-21; First posted 2017-06-19 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Joint Infection
Keywords: probabilistic antibiotherapy; prosthetic joint infection; treatment failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to establish a bacterial epidemiology in patients who present a prosthetic joint infection and for which a surgery is necessary. At the time of the first surgery, as the bacteria responsible for the infection are not known, a probabilistic antibiotherapy is initiated at once after the surgical treatment. The antibiotherapy is then adapted to the bacteria from samples collected during the surgery when they are identified (the delay is 14-21 days).

The study will focus on bacteria identified on samples collected during the surgery; the delay between the implantation of the prosthesis and the presentation of symptoms will be considered : more than one year vs. less than one year.

Investigators assume that there is not the same type of bacteria involved in those two cases of delays and that the probabilistic antibiotherapy may be not optimal when the symptoms are presented more than one year after implantation of the prosthesis. A probabilistic antibiotherapy not adapted lead to develop resistance for the bacteria and decrease the chance to cure the patient (increasing of relapse).

The result of this study will allow medical doctors to have an optimal probabilistic antibiotherapy, depending on the delay between implantation of the prosthesis and the presentation of the symptoms.

ELIGIBILITY:
Inclusion Criteria:

* patient with prosthetic joint infection and treated with probabilistic antibiotherapy, between 2010 and 2015, at the Croix-Rousse Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with prosthetic joint infection and treated with probabilistic antibiotherapy after a first surgery
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
identification of bacteria involved in patients with prosthetic joint infection | 3 weeks after the surgery
  The samples collected during the surgery are put in bacteriological culture media. Bacteriological culture of samples collected during surgery for all patients included is made allowing to identify which type of bacteria is involved in the infection, depending on the chronology of the infection (delay between implantation and the presentation of the symptoms [< 1 year vs. > 1 year])
collection of probabilistic antibiotic treatment in patients with prosthetic joint infection | the day of surgery
  The type of molecule used and dosage will be described. Probabilistic antibiotic treatment is initiated immediately after the surgery, before the bacteria is identified. The samples are put in bacteriological culture media. The time to obtain results is usually 3 weeks maximum after the surgery because this is the delay for slow-growing bacteria to grow. Then, the empirical treatment can be amended in order to have an antibiotic treatment adapted to the bacteria found.

SECONDARY OUTCOMES:
adverse events | up to 24 months after antibiotic therapy disruption
  This secondary outcome will focus on severe adverse events induced by this probabilistic antibiotherapy.
Treatment failure | up to 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- See also: Related Info — http://www.crioac-lyon.fr